CLINICAL TRIAL: NCT03613454
Title: Embolization in Splenic Trauma (ELSA)
Brief Title: Embolization in Splenic Trauma
Acronym: ELSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Andrew J. Gunn, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R18-097
Record Dates: First submitted 2018-07-12; First posted 2018-08-03 (Actual); Results first posted 2021-05-07 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Trauma to the Spleen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Splenic artery embolization with vascular embolic coils (Active Comparator)
  Interventions: Device: Splenic artery embolization with vascular embolic coils
- Splenic artery embolization with vascular embolic plugs (Active Comparator)
  Interventions: Device: Splenic artery embolization with vascular embolic plugs

INTERVENTIONS:
Device: Splenic artery embolization with vascular embolic coils — Splenic artery embolization with vascular embolic coils
  Arms: Splenic artery embolization with vascular embolic coils
Device: Splenic artery embolization with vascular embolic plugs — Splenic artery embolization with vascular embolic plugs
  Arms: Splenic artery embolization with vascular embolic plugs

SUMMARY:
Randomized, prospective, feasibility study to begin evaluating the efficacy, safety, and cost of using either coils or vascular plugs (VPs) for proximal splenic artery embolization in the setting of traumatic splenic injury.

DETAILED DESCRIPTION:
Splenic preservation rates are improved for participants with high-grade splenic injuries (defined as Grade III-V injuries by the American Association for the Surgery of Trauma (AAST) guidelines) when non-operative management is supplemented by image-guided, trans-catheter splenic artery embolization (SAE). SAE is currently the standard of care for hemodynamically stable participants with high-grade splenic injuries. In proximal SAE (pSAE), the mid-splenic artery is embolized between the origins of the dorsal pancreatic artery and pancreatica magna artery with either VPs or coils. This reduces the intra-splenic arterial pressure which allows the parenchyma time to heal. Splenic perfusion is maintained via a collateral pathway consisting of flow from the splenic artery proximal to the site of embolization through the smaller dorsal pancreatic artery to the transverse pancreatic artery to the pancreatica magna artery which then delivers a slower, smaller amount of blood to the splenic artery distal to the site of embolization. Additionally, collateral supply from the short gastric and gastroepiploic arteries helps to protect the spleen from infarction and/or abscess formation.

pSAE is most often accomplished using either coils or VPs as the embolic agent, both of which are FDA-approved and clinically-available. Coils have a long history of efficacy and safety for embolization and are thus familiar embolic agents to most endovascular specialists. Further, coils large enough to embolize the mid-splenic artery can be deployed through a standard micro-catheter, which means they can be used in even the most tortuous splenic arteries. However, multiple coils may need to be deployed in the same patient to achieve hemostasis in the mid-splenic artery that may increase their overall cost, iodinated contrast use, procedural time, and the radiation exposure to the participant and medical staff. Additionally, given the high-flow nature of the splenic artery, even an appropriately sized coil may migrate distally. A typical pSAE using coils will involve the deployment of one helical coil followed by multiple packing coils until hemostasis is achieved. VPs attempt to overcome the limitations of coils. For example, the deployment of a single VP can typically provide hemostasis in the mid-splenic artery which theoretically reduces procedural time, contrast load, and radiation exposure. Despite this, VPs are more expensive than coils on a per unit basis and are usually less familiar devices to endovascular specialists. Another drawback of VPs is that they cannot be deployed through a standard micro-catheter but rather require the advancement of a larger, stiffer 0.035 inch system into the mid-splenic artery. This may limit their use in very tortuous splenic arteries. Currently, the selection of embolic agent for pSAE is primarily based on operator experience and preference. The embolic efficacy, technical success, and cost of using coils compared to VPs has been evaluated in other diseases; yet, to the best of our knowledge, these embolic agents have never been compared for their use in pSAE, much less in a randomized, prospective fashion.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the University of Alabama at Birmingham (UAB) emergency room requiring embolization of the splenic artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-02-16 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Gunn, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- April Riddle, Harpersville, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Splenic Artery Embolization With Vascular Embolic Coils | Splenic Artery Embolization With Vascular Embolic Plugs
Started | 24 | 24
Completed | 23 | 23
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Splenic Artery Embolization With Vascular Embolic Coils | Splenic Artery Embolization With Vascular Embolic Plugs | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39 [26 to 61] | 34 [26 to 50] | 38 [26 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 18 | 17 | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Enrolled Within 18 Months of Study Initiation
Description: The primary outcome of the study will be enrolling 50 participants in the study within 18 months of study initiation with adequate 30 day follow-up on all participants.
Time Frame: Through study completion, an average of 1 year
Population: Two participants dropped out due to protocol violation (invalid consent)
Measure: Count of Participants; unit: Participants
Arm/Group | Splenic Artery Embolization With Vascular Embolic Coils | Splenic Artery Embolization With Vascular Embolic Plugs
Number analyzed (Participants) | 23 | 23
Participants | 23 | 23

2. Secondary Outcome: Number of Participants With Embolization Success
Description: This outcome will be measured by the ability of the operator to deploy the required embolic with resultant stasis in the splenic artery. This will be compared between the two groups.
Time Frame: Through study completion, an average of 1 year
Population: Two participants dropped out due to protocol violation (invalid consent)
Measure: Count of Participants; unit: Participants
Arm/Group | Splenic Artery Embolization With Vascular Embolic Coils | Splenic Artery Embolization With Vascular Embolic Plugs
Number analyzed (Participants) | 23 | 23
Participants | 22 | 20

3. Secondary Outcome: Number of Participants With Immediate Complications
Description: This outcome will be measured by the number of intra-procedural complications and compared between the two groups
Time Frame: During the embolization procedure, an average of 1 hour
Population: Two participants dropped out due to protocol violation (invalid consent)
Measure: Count of Participants; unit: Participants
Arm/Group | Splenic Artery Embolization With Vascular Embolic Coils | Splenic Artery Embolization With Vascular Embolic Plugs
Number analyzed (Participants) | 23 | 23
Participants | 2 | 1

4. Secondary Outcome: Number of Participants With Splenic Salvage
Description: This outcome will be measured by splenic salvage rate at 30 days and compared between groups. Splenic salvage was defined as the absence of splenectomy in the medical record or per patient report.
Time Frame: 30 days after procedure
Population: Two participants dropped out due to protocol violation (invalid consent)
Measure: Count of Participants; unit: Participants
Arm/Group | Splenic Artery Embolization With Vascular Embolic Coils | Splenic Artery Embolization With Vascular Embolic Plugs
Number analyzed (Participants) | 23 | 23
Participants | 22 | 23

5. Secondary Outcome: Radiation Exposure
Description: The radiation exposure during the embolization procedure for each embolic will be measured and compared.
Time Frame: During the embolization procedure, an average of 1 hour
Population: Two participants dropped out due to protocol violation (invalid consent)
Measure: Median (Inter-Quartile Range); unit: mGy
Arm/Group | Splenic Artery Embolization With Vascular Embolic Coils | Splenic Artery Embolization With Vascular Embolic Plugs
Number analyzed (Participants) | 23 | 23
mGy | 250 [172 to 671] | 380 [221 to 675]

6. Secondary Outcome: Contrast Volume
Description: The amount of contrast used during the procedure will be measured for each group and compared.
Time Frame: During the embolization procedure, an average of 1 hour
Population: Two participants dropped out due to protocol violation (invalid consent)
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Splenic Artery Embolization With Vascular Embolic Coils | Splenic Artery Embolization With Vascular Embolic Plugs
Number analyzed (Participants) | 23 | 23
mL | 54 [41 to 60] | 60 [50 to 75]

ADVERSE EVENTS:
Time Frame: Complications were recorded within 30 days from the procedure.
Description: Two participants dropped out due to protocol violation (invalid consent).
Arm/Group | Splenic Artery Embolization With Vascular Embolic Coils | Splenic Artery Embolization With Vascular Embolic Plugs
All-Cause Mortality (participants affected / at risk) | 1/23 | 1/23
Serious Adverse Events (participants affected / at risk) | 1/23 | 1/23
Other Adverse Events (participants affected / at risk) | 1/23 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Splenic Artery Embolization With Vascular Embolic Coils (N=23) | Splenic Artery Embolization With Vascular Embolic Plugs (N=23)
Coil migration (Surgical and medical procedures) | 1 (1) | 0 (0)
Vascular injury (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Splenic Artery Embolization With Vascular Embolic Coils (N=23) | Splenic Artery Embolization With Vascular Embolic Plugs (N=23)
Coil migration (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT03613454/Prot_SAP_000.pdf